CLINICAL TRIAL: NCT05196906
Title: The Clinical Outcomes Comparing the Modified Broström vs Anatomic Reconstruction Operation in Chronic Lateral Ankle Instability and Generalized Joint Laxity
Brief Title: The Clinical Outcomes of the Modified Broström vs Anatomic Reconstruction Operation in CLAI and GJL
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jiang Dong, Chief physician, Peking University Third Hospital
Other Study IDs: M2021565
Record Dates: First submitted 2021-12-27; First posted 2022-01-19 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-01

CONDITIONS: Ankle Sprains; Instability, Joint; Joint Hypermobility
Keywords: chronic lateral ankle instability; generalized joint laxity; re-injury; modified Brostrom operation; anatomic reconstruction
MeSH Terms: conditions — Ankle Injuries; Joint Instability; Reinjuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Modified Broström operation group: Patients who accept a modified Broström operation
  Interventions: Procedure: Modified Broström operation and anatomic reconstruction operation
- Anatomic reconstruction operation group: Patients who accept an anatomic reconstruction
  Interventions: Procedure: Modified Broström operation and anatomic reconstruction operation

INTERVENTIONS:
Procedure: Modified Broström operation and anatomic reconstruction operation — Patients with CLAI and GJL will accept the Modified Broström operation or anatomic reconstruction operation.

SUMMARY:
Investigators designed this prospective cohort study to compare the clinical outcomes of modified Broström operation and anatomical reconstruction for the treatment of CLAI and GJL.

DETAILED DESCRIPTION:
The modified Broström operation is still the first line to treat chronic lateral ligament instability (CLAI). However, some studies indicate the modified Broström operation may bring a higher rate of re-injury in generalized joint laxity (GJL). Anatomical reconstruction was reported to generate similar results and less rate of re-injury compared in patients with CLAI. However, the clinical outcomes of the two operations are not discussed in CLAI and GJL. So, investigators designed this prospective cohort study. The primary outcomes are Karlsson, Foot and Ankle Outcome Score (FAOS), and Foot and Ankle Ability Measure (FAAM) scores. The secondary outcomes are anterior displacement and talar tilt angle in stress radiography, the rate of re-injury.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of lateral ankle pain and instability Beighton score ≥4 Age with 18 to 60 years

Exclusion Criteria:

Patients with an acute or subacute ankle injury (within 3 months) Injury of the deltoid ligament Alignment of lower extremity greater than 5 degrees Fractures of the lower extremity Stage III or IV osteoarthritis Patients who refused to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients who go to visit a doctor for persistent lateral ankle pain and instability over three months and invalid conservative treatment, with the age of 16- 50 years. If the Beighton score of the patient is ≥4 and the exclusion criteria are met, he or she is going to be advised to participate in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Karlsson score | postoperative Karlsson score at 1 year.
  This score is a primary scale for lateral ankle instability
Karlsson score | postoperative Karlsson score at 2 years.
  This score is a primary scale for lateral ankle instability

SECONDARY OUTCOMES:
Anterior displacement and talar tilt angle in stress radiography | postoperative radiographic measures at 2 years.
  The outcomes are common indicators for evaluation the lateral stability of ankle

OTHER OUTCOMES:
Rate of re-injury | the rate of re-injury at 2 years.
  After surgery, the rate of patients re-sprain
Signal to noise value of the anterior talofibular ligament | 6 months post-treatment
  Signal to noise value of the anterior talofibular ligament
Signal to noise value of the anterior talofibular ligament | 12 months post-treatment
  Signal to noise value of the anterior talofibular ligament
Signal to noise value of the anterior talofibular ligament | 2 years post-treatment
  Signal to noise value of the anterior talofibular ligament

CONTACTS AND LOCATIONS:
Overall Officials: Dong Jiang, MD, Principal Investigator — Peking University Third Hosptial
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The demographics data, Beighton score, primary and secondary outcomes would be available to other researchers

REFERENCES:
- [Background] de Vries JS, Krips R, Sierevelt IN, Blankevoort L, van Dijk CN. Interventions for treating chronic ankle instability. Cochrane Database Syst Rev. 2011 Aug 10;(8):CD004124. doi: 10.1002/14651858.CD004124.pub3. PMID 21833947
- [Background] Michels F, Cordier G, Guillo S, Stockmans F; ESKKA-AFAS Ankle Instability Group. Endoscopic Ankle Lateral Ligament Graft Anatomic Reconstruction. Foot Ankle Clin. 2016 Sep;21(3):665-80. doi: 10.1016/j.fcl.2016.04.010. PMID 27524711
- [Background] Sacks HA, Prabhakar P, Wessel LE, Hettler J, Strickland SM, Potter HG, Fufa DT. Generalized Joint Laxity in Orthopaedic Patients: Clinical Manifestations, Radiographic Correlates, and Management. J Bone Joint Surg Am. 2019 Mar 20;101(6):558-566. doi: 10.2106/JBJS.18.00458. No abstract available. PMID 30893238
- [Background] Xu HX, Lee KB. Modified Brostrom Procedure for Chronic Lateral Ankle Instability in Patients With Generalized Joint Laxity. Am J Sports Med. 2016 Dec;44(12):3152-3157. doi: 10.1177/0363546516657816. Epub 2016 Aug 5. PMID 27496909
- [Background] Park KH, Lee JW, Suh JW, Shin MH, Choi WJ. Generalized Ligamentous Laxity Is an Independent Predictor of Poor Outcomes After the Modified Brostrom Procedure for Chronic Lateral Ankle Instability. Am J Sports Med. 2016 Nov;44(11):2975-2983. doi: 10.1177/0363546516656183. Epub 2016 Aug 1. PMID 27480980